CLINICAL TRIAL: NCT05865899
Title: Impact of High Tibial Osteotomy in Preventing Disease Progression in Medial Knee Osteoarthritis: Quantifying the Effects on Cartilage and Subchondral Bone by Using a Combined Biomechanical and Medical Imaging Approach.
Brief Title: Impact of High Tibial Osteotomy in Preventing Degenerative Disease Progression in Medial Knee Osteoarthritis.
Acronym: HTO-IOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-2018-12368274
Record Dates: First submitted 2023-03-23; First posted 2023-05-19 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis; Cartilage Degeneration; Malalignment, Bone
Keywords: Knee; Osteoarthritis; Varus; Malalignment; Cartilage; Correction Accuracy
MeSH Terms: conditions — Osteoarthritis, Knee; Bone Malalignment; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgical (Experimental): patients who undergo high tibial osteotomy procedure
  Interventions: Procedure: valgus producing medial opening wedge high tibial osteotomy
- conservative (No Intervention): patients who undergo conservative treatment

INTERVENTIONS:
Procedure: valgus producing medial opening wedge high tibial osteotomy — Valgus producing Opening wedge high tibial osteotomy will be performed through a medial incision at the proximal tibia and stabilized with a plate and screws. Hardware will be removed within 10-12 months to avoid soft tissue irritation.
  Arms: surgical

SUMMARY:
High tibial osteotomy (HTO) surgical procedure can lead to clinically significant improvements in the cartilage and in subchondral bone quality, with a slow down of the osteoarthritis (OA) progression.

Aim of the project is to:

(i) clinically validate a 3D planned HTO surgical approach, through a quantitative grading of OA progression in a prospective randomized case-control clinical trial; (ii) correlate the internal knee loads with the changes assessed in cartilage and subchondral bone status to verify the hypothesis that HTO induced mechanical changes are associated with clinically significant OA improvements; (iii) relate imaging data with cartilage and subchondral bone mechanical properties, in order to classify OA progression in a more sensitive manner and allow a more precise diagnosis of the pathology stage.

DETAILED DESCRIPTION:
High tibial osteotomy (HTO) is a well tracked procedure aimed to reduce the overload in the medial compartment of the varus knee with early and mid-stage osteoarthritits (OA).

Clear evidence still lacks regarding whether it has the ability to determine regenerative processes in the cartilage and subchondral bone. Furthermore, prospective randomised analysis regarding the effectiveness of HTO with respect to conservative treatment are needed.

The hypothesis is that an accurately planned HTO surgery result in measurable changes in the internal knee biomechanics, leading to clinically significant improvements in cartilage and subchondral bone quality, slowing down OA progression.

Accurate HTO could thus become the first choice in young/fit patients with medial knee OA, preserving their bone stock, slowing down OA progression and eventually reversing its trend, with a high impact on patients' quality of life and on public health system spending.

Aims of the study:

1. To quantify by quantitative imaging and subject-specific modeling the biomechanical changes induced in patients' joint by accurate HTO surgery, and the consequent changes of articular tissues composition and structure, related to OA progression.
2. To evaluate the surgical accuracy of a new 3D HTO planning system. Once association of biomechanical corrections with clinical outcome is established (Aim 1), such 3D HTO planning will help surgeons performing personalized HTO corrections.
3. To define an enhanced methodology for OA staging, by correlating quantitative medical imaging with mechanical properties of cartilage and subchondral bone.

Metodologies and statistical analyses:

Sample Size:The primary outcome of the study is the clinical assessment of cartilage/subchondral bone. In absence of standard subchondral bone scores, sample size has been determined on MRI T2 relaxometry, a reliable quantitative descriptor of cartilage in OA. Power analysis, based on cartilage T2 variations due to HTO (Independent t test, T2 expected difference 3.5 ms, standard deviation 4.5 ms, significance level 0.05, power 0.8, one tail), indicated 44 patients (22 per group). We target to enroll 50 patients to compensate for possible drop-outs.

Surgical technique: opening wedge HTO will be performed through a medial incision and stabilized with a plate and screws. Hardware will be removed within 10-12 months to avoid soft tissue irritation.

Imaging assessment: cartilage morphology and composition will be assessed via T1rho and T2 mapping from 3T MRI. Subchondral bone density and orientation will be computed from CBCT images. To quantify the biomechanical changes induced by HTO, subject-specific musculoskeletal models of the lower limbs will be created from MRI with nmsBuilder freeware, and used to calculate (with OpenSim software) knee loads during daily motor activities from marker trajectories and ground reaction forces measured in the gait analysis. A knee joint model enabling calculation of cartilage contact pressure will be implemented. Arthroscopic assessment of cartilage will follow the International Cartilage Repair Society (ICRS) score. Histological analysis of cartilage biopsies will be performed.

ELIGIBILITY:
Inclusion Criteria:

* medial knee osteoarthritis in varus knee malalignment (> 4°)

Exclusion Criteria:

* Inability to sign informed consent
* joint infection
* inflammatory chronic disease
* previous major surgical procedure of the indexed knee (simple arthroscopy or meniscectomy would be not considered major procedure)
* BMI > 30

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Cartilage morphology and composition assessment via T1rho and T2 mapping from 3Tesla (3T) magnetic resonance imaging(MRI). | 3 years
  Baseline and one-year follow-up cartilage status will be assessed in order to detect changes in cartilage status after the treatment. Quantitative cartilage assessment will be perfomed using T1rho and T2 mapping sequences which will be gathered during MRI.
Subchondral bone morphological and structural analysis via Cone Bean Computed Tomography (CBCT) of the knee. | 3 years
  Baseline and one-year follow-up subchondral bone morphological and structural features will be assessed via CBCT analysis, which allow to perform a weight-bearing assessment of the knee bone status and morphology.
Clinical Score for Knee function 1 | 3 years
  Marx Activity Rating Scale (MARS) score is an outcome reporting measure to evaluate the activity level of patients with various knee disorders who participate in sports. The MARS focuses on four activity points: running, deceleration, cutting (changing directions while running) and pivoting. MARS form will be assessed at baseline, six-months and 1-year follow-up. Higher scores mean a better outcome, lower scores mean a worse outcome.
Clinical Score for Knee function 2 | 3 years
  The Knee Injury and Osteoarthritis Outcome score KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. The KOOS meets basic criteria of outcome measures and can be used to evaluate the course of knee injury and treatment outcome. KOOS form will be assessed at baseline, six-months and 1-year follow-up. Higher scores mean a better outcome, lower scores mean a worse outcome.
Clinical Score for Knee function 3 | 3 years
  IKDC Subjective and objective Knee Evaluation Form. The entire IKDC form, which includes a demographic form, current health assessment form, subjective knee evaluation form, knee history form, surgical documentation form, and knee examination form, may be used as separate forms. IKDC evaluation form will be assessed at baseline, six-months and 1-year follow-up. Higher scores mean a better outcome, lower scores mean a worse outcome.

SECONDARY OUTCOMES:
Gait analysis assessment | 3 years
  Gait analysis will be assessed at baseline and at one-year follow-up in order to detect changes in gait pattern after the treatment. The active movements will be assessed by gait analysis tracking systems to quantify gait pattern.
Scores for general health | 3 years
  Short- form survey (SF-12) is composed by two summary scores: a mental component score (MCS-12) and a physical component score (PCS-12). Higher scores mean a better outcome, lower scores mean a worse outcome.
Scores for pain | 3 years
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

CONTACTS AND LOCATIONS:
Locations (1):
- Stefano Zaffagnini, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No